CLINICAL TRIAL: NCT05607082
Title: COVID-19 Bivalent Booster Megastudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 851911
Record Dates: First submitted 2022-11-03; First posted 2022-11-07 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19 vaccination; behavioral science interventions; vaccination promotion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the different arms.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: As treated participants will receive text messages, there is no scope for blinding. Care providers will not be made aware of subjects' participation in the study, or assigned treatment arms. The study team will only receive data on subjects' assigned arms and outcomes at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Holdout control condition with no message (No Intervention): Participants will only receive the standard pharmacy messaging.
- Control condition with "waiting for you" message (Experimental): This control condition will use the text message that we've found to be the best performing in our last mega-study of vaccine text messages to recommend a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Control condition with "waiting for you" message with a GIF (Experimental): This control condition will use the text message that we've found to be the best performing in our last mega-study of vaccine text messages and includes a GIF to recommend a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Planning message recommending same time/location as last vaccination (Experimental): This condition will use a text message recommending the same time and location as the participant's last vaccination to get a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message from local pharmacy team (Experimental): This condition will use a text message from the participant's local pharmacist recommending a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message including link to resources combating misinformation (Experimental): This condition will use a text message including a link to to resources combating misinformation and then recommend a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message including link to resources combating misinformation with a GIF (Experimental): This condition will use a text message including a link to to resources combating misinformation and then recommend a COVID vaccination and will include a GIF.
  Interventions: Behavioral: COVID Booster text messages
- Message offering free round trip ride to the pharmacy (Experimental): This condition will use a text message offering a free round trip ride to the pharmacy to get a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message communicating latest data on COVID transmission in patient's area (Experimental): This condition will use a text message informing the participant of the latest data on COVID transmission in participant's area and recommend a COVID vaccination.
  Interventions: Behavioral: COVID Booster text messages
- Message encouraging vaccination in preparation for the holidays (Experimental): This condition will use a text message to encourage a COVID vaccination in preparation for the holidays.
  Interventions: Behavioral: COVID Booster text messages
- Message conveying the CDC recommends vaccination (Experimental): This condition will use a text message to encourage a COVID vaccination by conveying the CDC recommends vaccination.
  Interventions: Behavioral: COVID Booster text messages

INTERVENTIONS:
Behavioral: COVID Booster text messages — Participants will receive text messages per descriptions listed in the arms.
  Arms: Control condition with "waiting for you" message; Control condition with "waiting for you" message with a GIF; Message communicating latest data on COVID transmission in patient's area; Message conveying the CDC recommends vaccination; Message encouraging vaccination in preparation for the holidays; Message from local pharmacy team; Message including link to resources combating misinformation; Message including link to resources combating misinformation with a GIF; Message offering free round trip ride to the pharmacy; Planning message recommending same time/location as last vaccination

SUMMARY:
This megastudy is a massive randomized controlled trial. By randomizing participants to 10 different intervention conditions simultaneously, the investigators will be able to compare the effectiveness of different interventions to one another and to a control group (in which individuals will only receive the usual communications from their partner organization) to identify which interventions significantly increase vaccination rates. Pharmacy customers will be randomly assigned to receive one of the interventions designed by team scientists to encourage vaccination or to a control group. The baseline intervention will be based on the top-performing SMS intervention identified in the investigators previous megastudies on encouraging vaccination (Milkman et al., 2021b, 2022). Pharmacy customers will receive SMS messages conveying that a COVID booster vaccine is reserved or waiting for them at the pharmacy. Additional behavioral science messaging strategies will be tested by building off of this baseline intervention.

ELIGIBILITY:
Inclusion Criteria:

• Patient of a large retail pharmacy that has opted into receving SMS messages from the pharmacy and has received their primary COVID vaccination series.

Exclusion Criteria:

* The patient unsubscribed from texts before the send date and time of the patient's SMS/MMS message
* The patient received a bivalent COVID booster before the send date and time of the patient's SMS/MMS message.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2600000 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Patient uptake of the COVID bivalent booster | During the 30 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question

SECONDARY OUTCOMES:
Patient uptake of the COVID bivalent booster | 60 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question
Patient uptake of the COVID bivalent booster | 90 days after receiving the SMS/MMS intervention
  Whether patients receive a bivalent COVID booster at the pharmacy in question

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No